CLINICAL TRIAL: NCT01437878
Title: A Phase 2, Multi-center, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of Inhaled Iloprost on Endurance Time During Cardiopulmonary Exercise Testing in Patients With Pulmonary Hypertension Secondary to Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Ventavis in Patients With Pulmonary Hypertension (PH) Secondary to Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-063B201
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
Keywords: PH; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iloprost (Experimental): single dose inhalation using the power disc-6 with I-neb Adaptive Aerosol Delivery (AAD) system
  Interventions: Drug: Iloprost
- placebo (Placebo Comparator): matching placebo using the power disc-6 with I-neb AAD system
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloprost — 5ug dose of inhaled iloprost (20ug/mL solution) administered 6 to 9 times per day for 4 weeks
  Other Names: Ventavis
  Arms: iloprost
Drug: Placebo — matching placebo
  Arms: placebo

SUMMARY:
This is a phase 2, Multi-center, double-blind, randomized, placebo-controlled study to evaluate the effects of inhaled Iloprost in patients with pulmonary hypertension secondary to COPD. The main objective is to investigate the effect of iloprost on exercise endurance time during constant work rate cardiopulmonary exercise testing. Other efficacy and safety endpoints will additionally be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure
2. Male or female ≥ 40 and ≤ 75 years of age
3. Women of childbearing potential1 must use a reliable method of contraception
4. Clinical diagnosis of moderate to severe COPD, with an obstructive pattern on pulmonary function tests
5. Current or past smokers of ≥ 10 pack years
6. Ability to perform exercise testing without supplemental oxygen (in the best opinion of the investigator)
7. Confirmed pulmonary hypertension by right heart catheterization (RHC)

Exclusion Criteria:

1. Other causes of pulmonary hypertension than COPD
2. BMI > 35 kg/m2
3. Conditions considered as contraindications for cardiopulmonary exercise testing (CPET) and/or inability to pedal on a cycle ergometer
4. Pregnant or nursing
5. Currently (within 30 days prior to RHC) taking specific pulmonary arterial hypertension (PAH) therapy (e.g., bosentan, ambrisentan, tadalafil, sildenafil, epoprostenol, treprostinil, iloprost, beraprost)
6. Participation in any other clinical trial, except observational, or receipt of an investigational product within 30 days prior to RHC visit
7. Known concomitant life-threatening disease with a life expectancy < 12 months
8. Known hypersensitivity to iloprost or any of the excipients of the drug formulations

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Bodin, MD, Study Director — Actelion
Locations (11):
- United States (9):
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Hopital d'adultes de Brabois, Vandœuvre-lès-Nancy, France
- Hospital Clinic i Provincial, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at 4 centres in the US, one centre in France, and one site in Spain. First patient, first visit was 1 March 2012 and last patient, last visit was 30 November 2012.
Pre-assignment Details: A total of 22 patients were screened for the study, of these 20 were not randomized because they did not meet the selection criteria.
Period: Overall Study
Arm/Group | Iloprost | Placebo
Started | 1 (Patient discontinued the study prior to initiation of study treatment) | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Iloprost: single dose inhalation using the power disc-6 with I-neb AAD system
  Iloprost: 5ug dose of inhaled iloprost (20ug/mL solution) administered 6 to 9 times per day for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Iloprost | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Number; unit: participants]
  Age 64 years | 1 | 0 | 1
  Age 74 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  France | 1 | 0 | 1
  United States | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Endurance Time
Description: Change from baseline to week 4 in endurance time during constant work rate exercise testing
Time Frame: Baseline to week 4
Population: The study was prematurely terminated as after 1 year it was not possible to identify a suitable number of patients who satisfied the selection criteria. Only 2 patients were randomized prior to the termination of the study, and 1 patient received a single dose of active treatment. Therefore, there are inadequate data to evaluate efficacy.
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events up to 24 hours post-end of treatment (EOT), approximately 4 weeks
Time Frame: Baseline up to 24 hours post-EOT, approximately 4 weeks
Population: Total population
Measure: Number; unit: participants
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

3. Secondary Outcome: Change in Systolic Pulmonary Arterial Pressure
Description: On Day 1 patients underwent acute hemodynamic testing prior to and immediately after (no more than 15 minutes) the first dose of inhaled iloprost or placebo. All hemodynamic variables were measured using a Swan-Ganz catheter.
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Diastolic Pulmonary Arterial Pressure
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Mean Pulmonary Arterial Pressure
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Mean Right Atrial Pressure
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Cardiac Output
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Right Ventricular Pressure
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Pulmonary Vascular Resistance
Description: as for outcome 3
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in End Tidal Partial Pressure of Carbon Dioxide
Description: Change from baseline to week 4. Pulmonary gas exchange was measured during incremental and constant work rate exercise testing.
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in End Tidal Partial Pressure of Oxygen
Description: as for outcome 10
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Oxygen Uptake
Description: as for outcome 10
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Carbon Dioxide Output
Description: as for outcome 10
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Oxygen Uptake Per Heartbeat
Description: as for outcome 10
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Heart Rate
Description: Change from baseline to week 4. Heart rate was measured during incremental and constant work rate exercise testing.
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in Arterial Oxygen Saturation as Indicated by Pulse Oximetry
Description: Change from baseline to week 4. Arterial oxygen was determined by pulse oximetry during incremental and constant work rate exercise testing.
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in Tidal Volume
Description: Change from baseline to week 4. Tidal volume was measured during incremental and constant work rate exercise testing.
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in Minute Ventilation
Description: Change from baseline to week 4. Minute ventilation was measured during incremental and constant work rate exercise testing.
Time Frame: Baseline to week 4
Population: as for outcome 1
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 hours post-end of treatment
Description: Treatment-emergent adverse events
Arm/Group | Iloprost | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other